CLINICAL TRIAL: NCT00460902
Title: Evaluation of the H-Coil Transcranial Magnetic Stimulation(TMS) Device- Augmentation for Drug Resistant Depression
Brief Title: Evaluation of the Deep TMS H-Coil in the Treatment of Major Depression- Augmentation of Antidepressant Medication
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Moshe Isserles, MD, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 395/3.11.06(HMO)
Record Dates: First submitted 2007-04-15; First posted 2007-04-17 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Major Depression
Keywords: TMS; drug resistant depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Deep TMS stimulation (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- DTMS with positive cognitive-emotional provocation (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- DTMS with negative cognitive-emotional provocation (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS)

SUMMARY:
Evaluation of the novel deep TMS H-Coil design as an augmentation measure in the treatment of medication resistant major depression. Stimulation is administered with and without cognitive-emotional provocation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as suffering from treatment resistant major depression
* Right laterality

Exclusion Criteria:

* other major axis I diagnosis
* severe axis II diagnosis
* risk factors to convulsions
* history of drug abuse in the past year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
HAMILTON RATING SCALE FOR DEPRESSION 24 items | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Isserles, MD, MSc, Principal Investigator — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Beer Yaacov Medical Center, Beer Yaacov
  - Biological psychiatry unit, Psychiatric ward, Hadassah Medical organization, Jerusalem

REFERENCES:
- [Background] Isserles M, Rosenberg O, Dannon P, Levkovitz Y, Kotler M, Deutsch F, Lerer B, Zangen A. Cognitive-emotional reactivation during deep transcranial magnetic stimulation over the prefrontal cortex of depressive patients affects antidepressant outcome. J Affect Disord. 2011 Feb;128(3):235-42. doi: 10.1016/j.jad.2010.06.038. Epub 2010 Jul 21. PMID 20663568